CLINICAL TRIAL: NCT04898556
Title: Clinical Study to Evaluate the Efficacy of Prasterone Treatment for Atrophy Vulvovaginal in Postmenopausal Women With Vulvar / Vestibular Pain
Acronym: ROSA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Santiago Palacios (Other)
Responsible Party: Sponsor-Investigator, Dr. Santiago Palacios, Investigador Principal, Instituto Palacios
Organization: Instituto Palacios (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-ROSA2020; 2020-004517-12 (EudraCT Number)
Record Dates: First submitted 2021-02-09; First posted 2021-05-24 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vultar/vestibular pain; Dyspareunia; Vaginal dryness
MeSH Terms: conditions — Dyspareunia | interventions — Dehydroepiandrosterone; Control Groups

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, open, randomized and controlled clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): Patients who will undergo treatment with Intrarosa (Prasterone 6.5mg) in ovules, will apply one ovule a day before going to bed for 12 weeks.
  Interventions: Drug: Prasterone 6.5 MG
- Control Group (Placebo Comparator): Patients who will not undergo any treatment for vulvovaginal atrophy for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prasterone 6.5 MG — The dose to be applied will be one Intrarosa ovule (Prasterone 6.5mg) a day before going to bed for 12 weeks.
  Other Names: Active Treatment
  Arms: Active Treatment
Other: Placebo — Patients with a diagnosis of VVA who will not undergo treatment for 12 weeks.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
A prospective, open, randomized and controlled clinical intervention study in women over 45 years of age with a diagnosis of vulvovaginal atrophy (dryness and / or dyspareunia, etc.) and vulvar and / or vestibular pain. The efficacy of Prasterone treatment is evaluated in those patients willing to undergo the treatment compared to the control group.

DETAILED DESCRIPTION:
A sample of 50 women over 45 years of age with at least one year of amenorrhea and who require treatment for vulvovaginal atrophy of moderate and / or severe intensity and who present vulvar and vaginal pain within these symptoms will be chosen.

At the beginning of the study, after passing the selection criteria and signing the informed consent, the patients will be randomly assigned to one of the two arms of the study, (active group) or (control group), said assignment will be made randomly. Through a computer program where one or the other arm of treatment will be assigned to the patient at random to guarantee the homogeneity of both study groups and thus avoid selection biases.

ELIGIBILITY:
Inclusion Criteria:

* Women over 45 years of age with at least one year of amenorrhea and at least one symptom of vulvovaginal atrophy of moderate and / or severe intensity.
* Women with moderate to severe vulvar / vestibular pain
* Women without symptoms or signs of acute vaginal infection.
* Women without symptoms of urinary infection and a negative urine strip result.
* Woman willing to carry out the study procedures and comply with the visits.
* Woman who signs the Informed Consent.

Exclusion Criteria:

* Hormone treatment in the last three months for vulvovaginal atrophy
* Treatment with vaginal moisturizers in the last week for vulvovaginal atrophy
* Laser treatment in the last 6 months.
* Acute and recurrent urinary tract infections in the last 3 months.
* Acute genital infections (herpes, candida, etc)
* Personal history of cancer at any level
* Present alterations in the area to be treated, such as lacerations, abrasions or ulcers (resolution time at the medical discretion)
* Decompensated non-communicable chronic diseases (Diabetes Mellitus, Heart Disease ...)
* Participation in a clinical study 3 months before inclusion or during this study.
* Hypersensitivity to the active principle or any of the excipients
* Undiagnosed vaginal bleeding.
* Untreated endometrial hyperplasia
* Acute liver disease or a history of liver disease while liver function tests remain impaired.
* Current diagnosis or history of venous thromboembolism (deep vein thrombosis, pulmonary embolism)
* Known thrombophilic disorders (protein C, protein S, or antithrombin deficiency)
* Current or recent diagnosis of arterial thromboembolic disease (angina, myocardial infarction)
* Porphyria

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment for vulvar / vestibular pain for patients with vulvovaginal atrophy | Screening Visit 1 (Day 0)
  Clinical study to evaluate the efficacy of Prasterone treatment for vulvovaginal atrophy in postmenopausal women with vulvar / vestibular pain.
Treatment for vulvar / vestibular pain for patients with vulvovaginal atrophy | Visit 2 (Week 4)
  Clinical study to evaluate the efficacy of Prasterone treatment for vulvovaginal atrophy in postmenopausal women with vulvar / vestibular pain.
Treatment for vulvar / vestibular pain for patients with vulvovaginal atrophy | Visit 3 (Week 12)
  Clinical study to evaluate the efficacy of Prasterone treatment for vulvovaginal atrophy in postmenopausal women with vulvar / vestibular pain.

SECONDARY OUTCOMES:
Evaluation of vulvo vestibular pain | Screening Visit 1 (Day 0); Visit 2 (Week 4); Visit 3 (Week 12)
  Through the visual analog scale (VAS)
Evaluation of vulvovaginal vascularization | Screening visit 1 (Day 0); Visit 3 (Week 12)
  Through the ECO DOPPLER
Evaluation of Ph and cytological maturity index | Screening Visit 1 (Day 0); Visit 3 (Week 12)
  On the lateral side of the vagina we take the Ph sample through a strip, and the cytological maturity is taken through a swab to take a sample from the cervical area.
Evaluation of the clinical index of vulvar and vaginal health | Screening Visit 1 (Day 0); Visit 3 (Week 12)
  It is carried out through a clinical parameter that takes into account humidity, hydration, elasticity, pH among others ...

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No